CLINICAL TRIAL: NCT06583044
Title: Bruxism Awareness and Self-assessment in Dental Clinical Students: A Questionnaire Study
Brief Title: Bruxism Awareness in Dental Students
Acronym: BADS
Status: Completed | Type: Observational
Sponsor: Abant Izzet Baysal University (Other)
Responsible Party: Principal Investigator, Tuğba ŞAHİN, Assistant professor, Abant Izzet Baysal University
Other Study IDs: AIBU-DH-TS-03
Record Dates: First submitted 2024-08-26; First posted 2024-09-03 (Actual); Last update posted 2024-09-03 (Actual); Status verified 2024-08

CONDITIONS: Bruxism
Keywords: awareness; bruxism; dental students; questionnaire
MeSH Terms: conditions — Bruxism | interventions — Surveys and Questionnaires

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Dentistry clinical student diagnosed with bruxism: This group includes dental clinical students diagnosed with bruxism.
  Interventions: Other: Questionnaire
- Dentistry clinical student without bruxism diagnosis: This group includes dental clinical students diagnosed without bruxism.
  Interventions: Other: Questionnaire

INTERVENTIONS:
Other: Questionnaire — It includes 33 questions measuring awareness and knowledge about bruxism.

SUMMARY:
Clinical students in the Faculty of Dentistry were diagnosed with bruxism according to the bruxism assessment consensus 2018. A total of 128 students with (64) and without (64) bruxism, were asked 33 questions about their knowledge and self-awareness about bruxism.

DETAILED DESCRIPTION:
This study included systemically healthy individuals aged 18 to 27. Intraoral and extraoral examinations were performed on 128 students with (64) and without bruxism (64), 4th and 5th-grade dental students at Bolu Abant İzzet Baysal University who met the inclusion criteria. The diagnosis of bruxism was based on the 2018 International Consensus and data collected through a validated 33-item questionnaire covering general information and bruxism awareness. The questionnaire included questions on bruxism's types, risk factors, symptoms, and impact on periodontal tissues, with multiple-choice responses. Statistical analyses were performed using IBM SPSS Statistics, and p<0.05 was accepted as statistical significance

ELIGIBILITY:
Inclusion Criteria:

* Systemically healthy individuals

Exclusion Criteria:

* Individuals with mental retardation,
* Individuals with suicidal tendencies,
* Individuals with dementia,
* Individuals with psychosis

Ages: 18 Years to 27 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: The study included 4th and 5th dental students.
Sampling Method: Non-Probability Sample
Enrollment: 128 (Actual)
Dates: Start 2024-06-05 (Actual); Primary Completion 2024-06-25 (Actual); Study Completion 2024-06-25 (Actual)

PRIMARY OUTCOMES:
Bruxism Awareness Survey | Baseline
  Determines how much information the participants have about bruxism diagnosis, symptoms, risk factors, and treatment methods. It consists of yes-no questions with two options. One is an answer.
Bruxism Knowledge Level Survey | Baseline
  Participants are assessed to determine the extent to which they can diagnose bruxism through self-assessment. It consists of 3 to 7 multiple-choice questions. One of the answers is the correct answer, and the assessment is based on this.

SECONDARY OUTCOMES:
Bruxism symptoms Survey | Baseline
  It includes information about whether the participants experience bruxism symptoms and the impact of these symptoms. It consists of 3 to 7 multiple-choice questions. One of the answers is the correct answer, and the assessment is based on this.
Treatment and Follow-up Survey | Baseline
  It includes questions about whether patients with bruxism are treated, what treatment methods are used, and whether there is an improvement in symptoms after treatment. It consists of 3 to 7 multiple-choice questions. One of the answers is the correct answer, and the assessment is based on this.

CONTACTS AND LOCATIONS:
Overall Officials: TUGBA SAHIN, Principal Investigator — Abant Izzet Baysal University
Locations (1):
- Bolu Abant İzzet Baysal University, Bolu, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Sahin T. Bruxism awareness and self-assessment in dental clinical students: a questionnaire-based study. BMC Oral Health. 2024 Oct 15;24(1):1223. doi: 10.1186/s12903-024-04997-x. PMID 39407206